CLINICAL TRIAL: NCT02218164
Title: A Phase 2 Study of Capecitabine or 5-FU With Pegylated Interferon Alpha-2b in Unresectable/Metastatic Cutaneous Squamous Cell Carcinoma
Brief Title: Capecitabine or 5-FU With Pegylated Interferon Alpha-2b in Unresectable/Metastatic Cutaneous Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17759
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Squamous Cell Carcinoma of Skin; Carcinoma, Squamous Cell
Keywords: metastatic; cutaneous; skin cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Neoplasm Metastasis; Skin Neoplasms | interventions — peginterferon alfa-2b; peginterferon alfa-2a; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine or 5-FU with Pegylated Interferon alpha-2b (Experimental): Participants will start the Capecitabine pills on day 1 thru day 14 and be off for 7 days (day 15-day 21).
  Participants will receive 5-FU days 1-4 of each 21 day cycle.
  Participants will receive the Interferon alpha-2b injection weekly every week. The three week period is referred to as one cycle.
  After three cycles, new imaging studies will be performed that will measure how the disease is responding to treatment. Participants whose disease is stable or improved will undergo an additional 3 cycles of therapy and the imaging studies will be repeated. Again, participants whose disease is stable or improved will undergo a final 3 cycles of treatment (a total 27 weeks of treatment).
  Interventions: Drug: Pegylated Interferon alpha-2b; Drug: Capecitabine; Drug: 5-FU

INTERVENTIONS:
Drug: Pegylated Interferon alpha-2b — Drug administration will occur on an outpatient basis at the infusion center at Moffitt Cancer Center. Dose will be weight-based. Starting treatment doses of 3 mcg/kg will be given subcutaneously (SC) injection in the thigh, abdominal wall, or upper arm every week for a total of 27 weeks as tolerated.
  Other Names: PEG Interferon Alpha-2b; PEG-INTRON; PEGASYS
Drug: Capecitabine — Drug administration will be on an outpatient basis. Capecitabine will be administered at an initial dose of 800 mg/m^2 by mouth twice daily on days 1-14 of a 21 day cycle with days 15-21 off. This cycle will be repeated every 21 days during the study for a maximum of 9 cycles as tolerated. Administration via feeding tube in patients unable to swallow is permitted.
  Other Names: Xeloda
Drug: 5-FU — If participants are not able to acquire oral capecitabine, then treating physicians will start participants on infusional 5-FU which can be delivered via standard of care. Participants will need to have a port placed for continuous infusion treatments. 5-FU pumps will be activated in the infusion center at Moffitt Cancer Center with a starting dose of 800 mg/m^2 days 1-4, with pump removal on day 5 at the infusion center. 5-FU pumps will be attached every 21 days (1 cycle) for a maximum of 9 cycles.
  Other Names: 5-fluorouracil

SUMMARY:
The purpose of this study is to find out if the combination of two established anti-cancer therapies are beneficial in patients with squamous cell carcinoma of the skin. Specifically, investigators want to determine if the combination of 5-FU/Capecitabine (oral pills) and Interferon alpha-2b (injection) can help people with advanced cases of squamous cell carcinoma of the skin. For participants that are not approved for oral capecitabine, treating physicians will use continuous infusion 5-FU. Both 5-FU/Capecitabine and Interferon alpha-2b have been used separately to treat squamous cell carcinoma of the skin and are FDA approved in other cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed squamous cell carcinoma of the skin. Potential participants who present with "squamous cell carcinoma of unknown primary lesions" at the time of diagnosis will be eligible if patients have a plausible primary skin site removed in the past. Similarly, potential participants with neck, parotid, or facial lymph nodes positive for squamous cell carcinoma with no identifiable mucosal primary would also be eligible.
* Must have measurable disease, defined by Response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as at least one lesion that can be accurately measured in at least one dimension of >10 mm by CT, MRI, or calipers
* There is no limitation to prior treatments with local, regional, topical or systemic agents, except for prior systemic treatment with 5-fluorouracil or prodrugs thereof. Prior topical treatment with 5-fluorouracil is permitted. Patients who are on chronic daily doses of prednisone of greater than 10 mg are excluded. There is no restriction on timing of last treatments as long as patients have recovered from all expected toxicities and at least 21 days have passed since last administration.
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Karnofsky >=60%
* Must have normal organ and marrow function
* Must not be candidates for curative locoregional treatments. Patients with recurrent locoregional disease following surgery and/or radiation for who a resection is unacceptably morbid and unlikely to be curative are eligible.
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have had chemotherapy or radiotherapy within 21 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* May not be receiving any other investigational agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to either 5-FU/Capecitabine or Interferon
* Uncontrolled, ongoing illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or breastfeeding
* Any heart or lung transplant patient on immunosuppressive agents. Renal transplant patients are allowed if patient is willing to reduce immunosuppressive agents and understand risk of rejection and possible need to return to dialysis. Patients with Chronic Lymphocytic Leukemia (CLL) or other hematologic malignancies are allowed as long as they meet other criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from August 2014 through May 2017.
Groups:
- Capecitabine or 5-FU With Pegylated Interferon Alpha-2b: Capecitabine pills on day 1 thru day 14 and be off for 7 days (day 15-day 21). 5-FU days 1-4 of each 21 day cycle. Interferon alpha-2b injection weekly every week. 3 week period is referred to as one cycle.
  After 3 cycles, new imaging studies will be performed to measure how the disease is responding to treatment. Participants whose disease is stable or improved will undergo an additional 3 cycles of therapy and the imaging studies will be repeated. Again, participants whose disease is stable or improved will undergo a final 3 cycles of treatment (a total 27 weeks of treatment).
Period: Overall Study
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 72 [63 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 8
  Black or African American | 0
  Asian | 0
  Hispanic or Latino | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR: Stable Disease (SD); Partial Response (PR); Complete Response (CR). Response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR: disappearance of all target lesions; PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 9 weeks per participant
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Number analyzed (Participants) | 8
Participants
  Stable Disease | 4
  Complete Response | 1
  Partial Response | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: Alive without RECIST progression. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 1 year
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Number analyzed (Participants) | 8
months | 11.3 [8.21 to NA] — Upper limit never crosses the 50% threshold on the Kaplan Meier curve.

3. Secondary Outcome: Overall Survival (OS)
Description: OS: The time from registration to death or date of last contact. Participants with overall survival at 1 year. Kaplan-Meier estimator will be utilized.
Time Frame: 1 year
Population: All participants who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Number analyzed (Participants) | 8
Participants
  Expired in less than a year | 4
  Alive at the end of the year | 2
  Had not completed survival follow-up at closeout | 2

4. Secondary Outcome: Occurence of Treatment Related Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent SAEs, overall and per Event Description.
Time Frame: 1 year
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
Number analyzed (Participants) | 8
Participants
  Any Related SAE | 1
  Dehydration | 1
  INR Increased | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b (N=8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Medication error (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
INR increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Neoplasms - Other, Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine or 5-FU With Pegylated Interferon Alpha-2b (N=8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Arm wound (non-lesion) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, New Skin cancer - different histology (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Finger cracking (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Stomatitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Failure to thrive (General disorders) | 2 (3)
Injection site reaction (General disorders) | 3 (4)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (4)
Fever (General disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (6)
Weight loss (Investigations) | 3 (6)
INR increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Infections and infestations - Other, Staph (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (4)
Hematoma (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cardiac disorders - Other, Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, Right eye edema (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02218164/Prot_SAP_000.pdf